CLINICAL TRIAL: NCT07386197
Title: The Effect of Sealer Type and Obturation Technique on Postoperative Pain of Root Canal Treated Teeth
Brief Title: The Effect of Sealer Type and Obturation Technique on Postoperative Pain
Acronym: pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 313/2021; Deanship of Research (Other: Jordan University of Science and Technology)
Record Dates: First submitted 2026-01-15; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Dental Pulp Necrosis
Keywords: Root canal treatment; Obturation; Sealer; Postoperative pain
MeSH Terms: conditions — Dental Pulp Necrosis; Bites and Stings; Pain, Postoperative | interventions — Root Canal Obturation

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned into four treatment methods
Who Masked: Participant
Masking Description: The patient is blinded to the type of treatment, the operator is partly blinded until the stage of filling material placement since blinding at this point is not possible due to material differences
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AH Plus resin sealer with cold lateral compaction (Active Comparator): Obturation using cold lateral condensation and resin sealer
  Interventions: Procedure: Obturation of root canals
- AH Plus with warm vertical compaction (Active Comparator): Obturation using warm vertical compaction and resin sealer
  Interventions: Procedure: Obturation of root canals
- TotalFill bioceramic sealer with single-cone technique (Active Comparator): Obturation with single cone and bioceramic sealer
  Interventions: Procedure: Obturation of root canals
- TotalFill HiFlow with warm vertical compaction (Active Comparator): Obturation with warm vertical compaction and bioceramic sealer
  Interventions: Procedure: Obturation of root canals

INTERVENTIONS:
Procedure: Obturation of root canals — filling of root canal using different materials of resin based or bioceramic based and cold lateral condensation or warm vertical condenstion techniques
  Other Names: Root canal filling with bioceramic sealers

SUMMARY:
Postoperative pain is an important consideration in endodontic treatment, and its incidence may be influenced by both obturation technique and sealer type. This study focused on molars to minimize anatomical variability and provide a consistent assessment of pain associated with different endodontic protocols.

This study aimed to evaluate the incidence and level of postoperative pain in molars treated with root canal therapy, in relation to the type of sealer and obturation technique used.

DETAILED DESCRIPTION:
One hundred and twenty patients (aged 18-60 years; 63 males, 57 females) requiring root canal treatment of mandibular or maxillary molars will be included. Only teeth with necrotic pulp and asymptomatic apical periodontitis or previously extirpated pulp are considered. Patients will be randomly assigned to one of four groups (30 patients each): Group A-AH Plus resin sealer with cold lateral compaction (AH-CLC); Group B-AH Plus with warm vertical compaction (AH-WVC); Group C-TotalFill bioceramic sealer with single-cone technique (TF-SC); Group D-TotalFill HiFlow with warm vertical compaction (TF-WVC). Postoperative pain will be self-recorded using the Visual Analog Scale (VAS) and Verbal Rating Scale (VRS) at 6 hours, 1 day, 2 days, 3 days, and 1 week after treatment. Completed forms will be collected when patients returned for permanent coronal restoration. Analgesic use was also recorded. Data will analyzed using one way ANOVA and Chi square tests.

ELIGIBILITY:
Inclusion Criteria:

1. both male and female patients within
2. The age of 18-60 years old who required root canal treatment
3. Either mandibular or maxillary molars with the diagnosis of either; necrotic pulp with asymptomatic apical periodontitis,
4. Teeth with pulp extirpated ( previously initiated root canal treatment) regardless of the periapical status

Exclusion Criteria:

1. Teeth diagnosed with irreversible pulpitis;
2. Teeth with intracanal abberations or mishaps such as perforations, transportation, severe ledging , broken instruments, apical resorption or open apices;
3. Teeth requiring posts;
4. Any patient on long term steroid or any other medical condition that requires long term analgesic.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Pain level after obturation of root canals | 6 hours, 1 day, 2 days, 3 days and 1 week
  The level of pain the patient will experience after obturation of the teeth using a visual analogue scale and a numerical scale from 0-10. Zero is the minimum and 10 is the maximum. The higher the score the worse it is, the best technique will have low scores of pain

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Alhiyasat, PhD, Study Chair — Jordan University of Science and Technology
Locations (1):
- Jordan university of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request from the study principal
Supporting Information: Study Protocol
Time Frame: After publication of the data and up to 5 years
Access Criteria: Request via email to the study chair
URL: https://www.just.edu.jo/Pages/Default.aspx